CLINICAL TRIAL: NCT05726344
Title: Lactulose vs. Polyethylene Glycol as Bowel Preparation for Colonoscopy in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clínicas Dr. Manuel Quintela (Other)
Responsible Party: Principal Investigator, Ignacio Moratorio, Principal Investigator, Hospital de Clínicas Dr. Manuel Quintela
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 7477252
Record Dates: First submitted 2023-01-18; First posted 2023-02-13 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Lactulose; Polyethylene Glycol; Bowel Preparation; Colonoscopy; Bisacodyl
MeSH Terms: interventions — Lactulose; Bisacodyl; Water; polyethylene glycol 3350

STUDY DESIGN:
Intervention Model Description: An analytical, experimental, prospective study, specifically a triple blind randomized clinical assay (endoscopist, researchers and statistician) in which a bowel preparation is compared for colonoscopy with lactulose vs. Polyethylene Glycol.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Triple blind (endoscopist, researchers and statistician) randomized clinical assay.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lactulose group (Experimental): Patients participating in the study shall go on with their usual diet prior to colonoscopy. Three days before avoid consuming fruits, vegetables, seeds and cereals. A low residue soft and liquid diet is allowed.
  The day before the study, the group receiving lactulose shall take 4 tablets of Bisacodyl (5 mg) the day before the study at 6pm. Then, at 8pm a bottle of 250 mL (162.5g lactulose) of lactulose shall be dissolved in 600 mL of water and all contents (850 mL) shall be taken in 2 hours. At 10pm they have to drink 2 liters still water.
  Interventions: Drug: Lactulose
- Polyethylene glycol group (Experimental): Patients participating in the study shall go on with their usual diet prior to colonoscopy. Three days before avoid consuming fruits, vegetables, seeds and cereals. A low residue soft and liquid diet is allowed.
  The day before the study, the group receiving polyethylene glycol (PEG) should take 4 tablets of Bisacodyl (5 mg) at 4pm. Then, at 6pm, 3 bottles of PEG (Polyethylene glycol 3350 60 g; sodium chloride 1.46 g; potassium chloride 745 mg; Sodium bicarbonate 1.68 g; anhydrous sodium sulfate 5.68 g; pineapple flavoring 483 mg) shall be dissolved in 3 liters of water (1 bottle per liter) and they shall take half the preparation, that is 1 liter and a half in 2 hours. At 10pm they shall take the remaining contents in 2 hours.
  Interventions: Drug: Polyethylene Glycol 3350

INTERVENTIONS:
Drug: Lactulose — 4 tablets of Bisacodyl (5 mg) + 250 mL (162.5g lactulose) of lactulose + 600 mL of water + 2 L of water
  Other Names: Bisacodyl 20 mg; Water 600 mL
  Arms: Lactulose group
Drug: Polyethylene Glycol 3350 — 4 tablets of Bisacodyl (5 mg) + 3 bottles Polyethylene Glycol 3350 (Polyethylene glycol 3350 60 g; sodium chloride 1.46 g; potassium chloride 745 mg; Sodium bicarbonate 1.68 g; anhydrous sodium sulfate 5.68 g; pineapple flavoring 483 mg) + 3 L of water
  Other Names: Bisacodyl 20 mg; Water 3 L
  Arms: Polyethylene glycol group

SUMMARY:
Colonoscopy is the gold standard in bowel assessment when there is suspicion of colon and rectum pathology. Bowel cleansing is necessary to ensure an optimal visualization of colonic mucosa, allowing this form of detection and removal of polyps. Nowadays international recommendations have multiple bowel preparations. There are differences among them regarding adherence, tolerance and adverse effects. Lactulose (LAC) is widely used in treating constipation. However, there are some randomized clinical assays using LAC as bowel preparation with excellent results according to bowel preparation and tolerance scales. Adherence to bowel preparation significantly affects the result in the endoscopic study.

Safety of polyethylene glycol (PEG) formulations has been validated in several studies, it presents little severe side effects and the advantage of its applicability to patients with several comorbidities (heart, liver and kidney without water deprivation). However, its main disadvantage lies in the need to ingest large amounts of liquid (3-4L), generating intolerance thereto in 15%-45% of patients.

Bowel cleansing preparation with PEG is widely used in clinical practice. Considering that according to international studies reporting better tolerance and adherence with LAC; it is suggested to compare the level of bowel preparation, tolerance and adherence between two groups with LAC and PEG.

ELIGIBILITY:
Inclusion Criteria:

- Patients over 18 years with no bowel surgical procedures

Exclusion Criteria:

* Patients willingly deciding not to enter into the study
* Pregnant women
* Patient with colonic resections and/or ileostomies
* Inflammatory bowel disease
* Colonic optimization by prior colonoscopy with poor preparation
* Suspected intestinal occlusion or perforation, intussusception
* Patient with melenas
* Oral iron intake in the past 10 days
* Emergency colonoscopy
* Hypersensitivity to any of the components comprised in preparations.
* Diabetics
* Chronic kidney disease in dialysis
* Uncorrected severe dystonias
* Severe psychiatric illness (schizophrenia)
* Low IQ to understand bowel preparation
* Severe constipation (< 1 weekly stool)
* Chronic diarrhea with high rate (≥ 4 daily evenly loose consistency stools for more than 4 weeks)
* Unbalanced heart diseases (ischemic cardiopathology, congestive heart failure, unstable angina, arrhythmias and untreatable high blood pressure)
* Ascites

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2023-02-10 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Compare lactulose vs. Polyethylene Glycol as bowel cleansing preparation for colonoscopy | 6 months
  Compare the level of bowel preparation (by Boston Bowel Preparation Scale) between two groups with lactulose and Polyethylene Glycol.
  The minimum and maximum value is 0 and 9, respectively. A proper preparation is consider a Boston Bowel Preparation Scale ≥ 2 scores in each colonic segment. Unsuitable preparation a Boston Bowel Preparation Scale < 2 scores in any of the segments.
  Score 0: is considered a segment of unprepared colon with mucosa that cannot be observed given the presence of solid stool which does not disappear after cleansing.
  Score 1: part of the colonic mucosa is observed; other areas cannot be suitably assessed given the presence of staining, residual matter and/or opaque liquid.
  Score 2: little remaining residual matter and small matter fragments which do not prevent correct visualization of colonic mucosa in said segment.
  Score 3: colonic mucosa which can be entirely observed with no residual matter nor small fragments of matter and opaque liquid.
Establish Boston Bowel Preparation Scale inter and intra-observer variability | 7 months
  Two researchers shall review the endoscopic study videos and they shall complete the Boston Bowel Preparation Scale inter-observer questionnaire. Results obtained by the endoscopist in charge of the study and the observers shall be compared so as to establish inter-observer variability. Researchers shall analyze one month later again all colonoscopies recorded thus establishing Boston Bowel Preparation Scale of each endoscopy. Then results previously established shall be compared so as to establish intra-observer variability.
  The minimum and maximum value is 0 and 9, respectively. A proper preparation is consider a Boston Bowel Preparation Scale ≥ 2 scores in each colonic segment. Unsuitable preparation a Boston Bowel Preparation Scale < 2 scores in any of the segments.

SECONDARY OUTCOMES:
Assess tolerance between lactulose and Polyethylene Glycol. | 6 months
  To assess tolerance it will be considered: good tolerance those patients with 3 or less symptoms with no major criterion; regular tolerance those patients with 4-5 symptoms, without major criterion and bad tolerance those patients with 6 or more symptoms or 1 or more major criteria.
Assess adherence between lactulose and Polyethylene Glycol. | 6 months
  To assess adherence it shall be assessed if the preparation was completed as well as the will to repeat the same preparation in the future.
Assess side effects between lactulose and Polyethylene Glycol. | 6 months
  To assess side effects of both preparations that will be considered: nausea, vomiting, abdominal pain or bloating, sickness, lipothymia, palpitations, precordial pain, insomnia, anal pain or burning, dry mouth, tinnitus, unpleasant taste.
Establish colonoscopy global adenoma detection rate with lactulose and Polyethylene Glycol. | 6 months
  It correspond to the number of adenomas/adenocarcinomas (histological diagnosis) divided by the total number of colonoscopies performed times 100.
Establish colonoscopy cecal intubation rate in with lactulose and Polyethylene Glycol. | 6 months
  It correspond to the number colonoscopies visualizing ileocecal valve divided by the total number of colonoscopies performed times 100.

CONTACTS AND LOCATIONS:
Overall Officials: IGNACIO MORATORIO, MD, Principal Investigator — HOSPITAL DE CLINICAS; MARIA B RUSSO, MD, Principal Investigator — HOSPITAL DE CLINICAS; FLORENCIA RODRIGUEZ, MD, Principal Investigator — HOSPITAL DE CLINICAS
Locations (1):
- Hospital de Clinicas, Montevideo, Uruguay

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, Statistical Analysis Plan and Informed Consent Form
Supporting Information: Study Protocol, SAP, ICF
Time Frame: ENDED THE TRIAL